CLINICAL TRIAL: NCT05413655
Title: A Phase 2, Randomized, Double Blind, Placebo-Controlled Study of Oral EX039 As Add-on to Acetylcholine Esterase Inhibitors in Subjects with Mild Alzheimer's Disease
Brief Title: A Study of Oral EX039 in Subjects with Mild Alzheimer's Disease
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Excelsior (Industry)
Collaborators: Formosa Biomedical Technology Corp. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EX-039-10701
Record Dates: First submitted 2022-03-14; First posted 2022-06-10 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- 1000 mg (Experimental): The recruited patient randomly assigned to this arm will take 1000 mg EX039 per day
  Interventions: Drug: EX039
- 750 mg (Experimental): The recruited patient randomly assigned to this arm will take 750 mg EX039 per day
  Interventions: Drug: EX039
- placebo (Placebo Comparator): The recruited patient randomly assigned to this arm will take placebo per day
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: EX039 — The dosage form of EX039 is the capsule for oral use
  Arms: 1000 mg; 750 mg
Drug: Placebo — The dosage form of Placebo is the capsule for oral use
  Arms: placebo

SUMMARY:
This is a phase 2, randomized, double-blind, placebo-controlled study of oral EX039 as add-on to Acetylcholine Esterase Inhibitors in subjects with mild Alzheimer's disease.

ELIGIBILITY:
Inclusion Criteria:

* Aged 50-80 years.
* Clinical diagnosis of probable mild Alzheimer disease dementia based on National Institute of Neurological and Communicative Disorders and Stroke and the Alzheimer's Disease and Related Disorders Association (NINCDS/ADRDA criteria, 2011)
* Last time (which must be within 3 months ) of Mini Mental State Exam (MMSE) between 10-26.
* Last time (which must be within 3 months) of Clinical Dementia Rating (CDR) score of 1.
* Physically healthy and all laboratory assessments (including hematology, chemistry, urinalysis and electrocardiograph) are within normal range or meet the following criteria:

  * AST, ALT level ≦ upper limit of normal
  * Creatine Kinase (CK) concentration more than 3 times upper limit of normal
  * Serum creatinine level ≦ upper limit of normal
  * HbA1c more than 8.0
* Complaints of subjective memory impairment and cognitive disturbances by patients themselves or caregivers, including memory loss and at least one of the following cognitive disturbances: language, perceptual skills, attention, constructive abilities, orientation, problem solving, functional abilities.
* Cognitive deficits caused impairment in social or occupational function.
* Disease progression with gradual and continued decline from a previous level of functioning.
* Female subjects must be of non-childbearing potential (greater than 1 year without menstrual period in the absence of hormone replacement therapy) or surgically sterile. If pre-menopausal or menopausal for 1 year or less, must have a negative pregnancy test and must not be lactating at screening visit. Female subjects of childbearing potential and who are sexually active are required to practice adequate methods of birth control. Male subjects who are sexually active will also be required to use an adequate form of birth control.
* Has sufficient education equivalent to elementary education to communicate effectively and were capable of completing the assessments of the study.

Exclusion Criteria:

* Having other causes of dementia.
* Having substantial concomitant cerebrovascular disease (defined by a history of a stroke

  / intracranial hemorrhage temporally related to the onset of worsening of cognitive impairment) per investigator judgement.
* Medical history of cancer (except for basal cell carcinoma) and/or treatment for cancer within the last 5 years.
* Medical history or diagnosis of any of the following symptomatic and unstable / uncontrolled conditions per investigator's judgement:

  * Uncontrolled cardiovascular illnesses such as chronic congestive heart failure (with or without edema), tachycardia, arrhythmias, uncontrolled hypertension.
  * Significant ischemic heart disease, myocardial infarction within the last two years and/or with residual angina, orthopnea, conduction defects (ECG), or any other clinical significant heart disease classified as New York Heart Association (NYHA) III or IV.
  * Significant gastrointestinal disorders (for example gastrointestinal bleeding within the last two years, malabsorption syndromes, post-gastrectomy, or active peptic ulcer disease).
  * Uncontrolled endocrine disease such as uncontrolled diabetes mellitus or hyperthyroidism.
  * Unstable/Uncontrolled major depression.
  * Has neurological disease (other than dementia of Alzheimer's type, such as: Lewy body dementia - primary diagnosis, Huntington's disease, Parkinson's Disease, encephalitis, epilepsy, vascular or multiinfarct dementia, stroke, congenital mental deficiency, multiple sclerosis).
  * Significant pulmonary disease predisposing to hypoxia.
  * Has major physical illnesses (e.g. brain tumor, craniocerebral trauma, thyroid disease)
* Any other psychiatric disorders such as schizophrenia, or mental retardation.
* Any suicidal actions in the past 2 years (per investigator judgement i.e. actual attempt, interrupted attempt, aborted attempt, or preparatory acts or behavior).
* Hachinski Ischemic Score > 4
* Significant history of drug dependence or abuse (including alcohol, as defined in Diagnostic and Statistical Manual of Mental Disorders [DSM-V] or in the opinion of the investigator)
* Clinically significant uncompensated hearing loss in the judgment of the investigator. Use of hearing aids is allowed.
* Has other condition(s) that in the opinions of investigators to be ineligible to participate in this study, e.g. Subject who cannot swallow the capsule whole.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-08-08 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Change in Alzheimer's Disease Assessment Scale-cognitive | Week 28
  Mean change from baseline in Alzheimer's Disease Assessment Scale-cognitive subscale measured at the end of week 28. Total scores range from 0-70, with higher scores (≥ 18) indicating greater cognitive impairment.
Change in Clinical Dementia Rating-Sum of Boxes | Week 28
  Mean change from baseline in Clinical Dementia Rating-Sum of Boxes (CDR-SB). measured at the end of week 28. Total scores range from 0 to 18, with higher scores indicating more worsening.

SECONDARY OUTCOMES:
Change in Clinician's Interview-Based Impression of Change Plus Caregiver Input | Week 4, 12, 20, 28
  Scorings of Clinician's Interview-Based Impression of Change Plus Caregiver Input (CIBIC-Plus) at the end of week 4, 12, 20, and 28.
Incidence of Treatment-Emergent Adverse Events | Week 30
  To assess the safety and tolerability of EX039
Responder rate assessment | Week 28
  The percentage of the recruited subjects whose mean change from baseline in Alzheimer's Disease Assessment Scale-cognitive subscale (ADAS-cog) measured at the end of week 28 is improved (≧4) without deterioration of CDR-SB and CIBIS-Plus

CONTACTS AND LOCATIONS:
Overall Officials: Ching-Kuan Liu, Dr., Principal Investigator — Kaohsiung Medical University
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No
There won't be any individual participant data shared to other researchers.